CLINICAL TRIAL: NCT01535144
Title: Comparative Study of Osteosynthesis for Chevron Osteotomy of Hallux Valgus Using Degradable Versus Non-degradable Metallic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syntellix AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: syn09-01
Record Dates: First submitted 2012-02-01; First posted 2012-02-17 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- degradable metallic device (Experimental)
  Interventions: Device: Fracture compressing screw ZfW 102 Königsee Implantate GmbH
- non-degradable metallic device (Active Comparator)
  Interventions: Device: Fracture compressing screw titanium Königsee Implantate GmbH

INTERVENTIONS:
Device: Fracture compressing screw ZfW 102 Königsee Implantate GmbH — Comparison of two metallic implantable fracture compressing screws
  Arms: degradable metallic device
Device: Fracture compressing screw titanium Königsee Implantate GmbH — Comparison of two metallic implantable fracture compressing screws
  Arms: non-degradable metallic device

SUMMARY:
The purpose of the study is to show the equivalence of a new degradable metallic device to a non-degradable metallic device in patients with Hallux Valgus.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with an age of 40 to 79 years at the day of surgery
* Symptomatic Hallux Valgus
* Radiological criterium area of proximal joint angle
* Normal motorically functions
* Female patients of childbearing age must be using two reliable contraception methods

Exclusion Criteria:

* Previous bone and/or soft tissue surgeries of the the first metatarsal of the respective foot
* BMI > 32
* Cysts of the first metatarsal of the respective foot
* Neurological disorders with modified motorically functions
* Clinical evidence of osteoporosis
* Chronic renal impairment
* Known hypersensitivity to components of the implants
* Regular administration of medications containing the metallic elements of the degradable implant
* Pregnant or lactating women
* Current participation in another clinical trial or within 30 days before surgery

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
difference of metatarsal angles in degree post surgery and 6 months after surgery | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Windhagen, Prof., MD, Principal Investigator — Clinic for Orthopaedic Surgery (in the Annastift Hospital)
Locations (1):
- Clinic for Orthopaedic Surgery (in the Annastift Hospital), Hanover, Lower Saxony, Germany